CLINICAL TRIAL: NCT03859544
Title: Molecular Prognosis of Lymphomas of the Central Nervous System (ALYCE-molecular)
Acronym: ALYCEmolecular
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL17_0692
Record Dates: First submitted 2019-02-28; First posted 2019-03-01 (Actual); Last update posted 2019-03-01 (Actual); Status verified 2019-02

CONDITIONS: Central Nervous System Lymphoma
MeSH Terms: interventions — Retrospective Studies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Retrospective study — Retrospective study to search mutations associated with Central nervous system lymphoma and study of the prognostic impact (overall survival and progression-free survival) of these mutations.

SUMMARY:
Central nervous system lymphoma (PCNSL) is a diffuse large B cell lymphoma (DLBCL) entity with a particularly poor prognosis (median survival less than 3 years). They are still poorly characterized biologically, largely because of their rarity (300 cases / year in France) and the difficulty for obtaining a material of sufficient quality and quantity. It is nevertheless assumed that their pathophysiology is particular, since they develop exclusively in an immunological sanctuary, and that they present some characteristic molecular abnormalities (mutation of MYD88 or TBL1XR1 for example).

A collection of 74 PCNSLs has created, clinically annotated, from which frozen material is available in addition to the material fixed and included in paraffin (cohort ALYCE). Informed consent was gathered for all patients. Comparative Genomic Hybridization-array analysis of this cohort has already revealed abnormalities associated with a poor prognosis (unpublished data). The objective of this study is to complete this analysis by sequencing a panel of 96 mutant genes recurrently in DLBCLs and PCNSLs, and the molecular determination of the original cell by the (RT-MLPA) Reverse Transcriptase-Multiplex Ligation-dependent Probe Amplification technique.

The integration of genetic, molecular and transcriptomic data may define prognostic markers and open perspectives for translational research in PCNSL.

ELIGIBILITY:
Inclusion Criteria:

* Adults
* With a lymphoma of the central nervous system
* Patients having signed the consent for the conservation of their samples within the cohort

Exclusion Criteria:

* <18 old years
* Other diagnosis than lymphoma of the central nervous system
* No consent form signed

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This study focuses on adult subjects (male and female) with central nervous system lymphoma.
Sampling Method: Non-Probability Sample
Enrollment: 74 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | Up to 48 months
  Analysis of progression-free survival correlated with genomic data and mutation data

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'hématologie biologique - Centre Hospitalier Lyon Sud - HCL, Pierre-Bénite, France

IPD SHARING:
Plan to Share IPD: No